CLINICAL TRIAL: NCT02296671
Title: Personalized Therapy for Esophagogastric Cancer Using Thymidylate Synthase Genetic Markers
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Was unable to accrue any patients
Sponsor: Washington University School of Medicine (Other)
Collaborators: Gateway for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201412051
Record Dates: First submitted 2014-11-18; First posted 2014-11-20 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Esophagogastric Cancer
MeSH Terms: interventions — Pemetrexed; Oxaliplatin; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PEMOX (Experimental): Pemetrexed will be given intravenously (IV) on an outpatient basis on Day 1 of each 14-day cycle over 10 minutes. Oxaliplatin will be given (IV) on an outpatient basis on Day 1 of each 14-day cycle at a dose over 120 minutes. Drugs may be given in either order.
  -Oxaliplatin will be administered on Day 2 for Cycle 1 only. **
  Interventions: Drug: Pemetrexed; Drug: Oxaliplatin; Genetic: Germline genotyping analyses for TSER
- FOLFOX (Experimental): The modified FOLFOX-6 regimen is the following drugs given every 14 days:
  * Oxaliplatin on Day 1 of each cycle
  * Leucovorin over 120 minutes on Day 1 of each cycle
  * 5-FU bolus and continuous infusion over 46 hours beginning on Day 1 of each cycle
    * Oxaliplatin will be administered on Day 2 for Cycle 1 only and the 5-FU infusion will be interrupted at 20 hours so that the FLT-PET scan can be performed (only for FLT-PET scan eligible patients).
  Interventions: Drug: Pemetrexed; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Genetic: Germline genotyping analyses for TSER

INTERVENTIONS:
Drug: Pemetrexed
  Other Names: Alimta®
Drug: Oxaliplatin
  Other Names: Eloxatin®
Drug: Leucovorin
  Other Names: Wellcovorin
  Arms: FOLFOX
Drug: Fluorouracil
  Other Names: 5FU; 5-Fluorouracil; Adrucil®
  Arms: FOLFOX
Genetic: Germline genotyping analyses for TSER

SUMMARY:
In this study the investigators aim to: 1) confirm the objective response rate (ORR) observed in the investigators initial study for patients with the TSER*2/*2 genotype 2) determine whether PEMOX regimen is more worthy of future development for this patient genotype selected population than FOLFOX based on the data indicating that pemetrexed may be a better TS targeted agent than 5-FU.

Patients who are homozygous for the TSER*2 allele (TSER*2/*2) will be able to continue in the study and will be randomized. Patients with other TSER genotypes will not be included and will be considered screen fails.

The first 8 patients with the TSER*2/*2 genotype will be randomized 1:1 to receive treatment with either PEMOX or FOLFOX (4 in each group).

Analysis of the objective response rate (ORR) in each treatment arm will occur after the first 8 patients are enrolled. Using the proposed Bayesian design, subsequent patients will be preferentially assigned to the "better performing" treatment arm based on continuous real-time reassessments of ORR results.

ELIGIBILITY:
Inclusion Criteria:

Pre-Registration Inclusion Criteria

* Histologically or cytologically confirmed unresectable or metastatic esophagogastric adenocarcinoma.
* Measurable disease defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as >10 mm with CT scan, as >20 mm by chest x-ray, or >10 mm with calipers by clinical exam. PET/CT scan is acceptable as a substitute for a CT scan if the CT portion of the PET/CT is of identical diagnostic quality to a diagnostic CT scan.
* At least 18 years of age.
* ECOG performance status < 2
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Registration Inclusion Criteria

* TSER genotype *2/*2
* ECOG performance status < 2
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,500 cells/mm3
  * Platelets ≥ 100,000 cells/mm3
  * Total bilirubin < 1.5 x IULN
  * AST(SGOT)/ALT(SGPT) < 3.0 x IULN
  * Creatinine within normal institutional limits OR Creatinine clearance ≥ 45 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.

Exclusion Criteria:

Pre-Registration Exclusion Criteria

* Prior therapy for this cancer.
* A history of other malignancy ≤ 5 years previous with the exception of basal cell or squamous cell carcinoma of the skin which were treated with local resection only or carcinoma in situ of the cervix.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known HIV-positivity on combination antiretroviral therapy because of the potential for pharmacokinetic interactions with pemetrexed and/or oxaliplatin. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Registration Exclusion Criteria

* Currently receiving any other investigational agents.
* Known brain metastases. Patients with known brain metastases must be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to pemetrexed, 5-FU, leucovorin or oxaliplatin, or other agents used for premedication in the study.
* Pregnant and/or breastfeeding. Patient must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2018-09 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline, end of every 4th cycle, and end of treatment (estimated average of 6 months)
  ORR=complete response + partial response by RECIST criteria
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Overall survival (OS) | Every 3 months for up to 4 years from the date of study registration or until death, whichever occurs first
  OS = The length of time from the start of treatment to time of death.
Quality of life | Baseline and Day 1 of each cycle through Cycle 5 Day 1 (approximately Day 70)
  Quality of life will be assessed by the EORTC QLQ-C30 and the EORTC QLQ-STO22

CONTACTS AND LOCATIONS:
Overall Officials: A. Craig Lockhart, M.D., Principal Investigator — Washington University School of Medicine

REFERENCES:
- [Background] Goff LW, Thakkar N, Du L, Chan E, Tan BR, Cardin DB, McLeod HL, Berlin JD, Zehnbauer B, Fournier C, Picus J, Wang-Gillam A, Lee W, Lockhart AC. Thymidylate synthase genotype-directed chemotherapy for patients with gastric and gastroesophageal junction cancers. PLoS One. 2014 Sep 18;9(9):e107424. doi: 10.1371/journal.pone.0107424. eCollection 2014. PMID 25232828
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu